CLINICAL TRIAL: NCT01246869
Title: Assessment of Primary and Metastatic Brain Tumor Hypoxia With 18F-Fluoromisonidazole, [18F]Fluoro-2-deoxy-D-glucose (FDG) and [15O]Water (H215O)
Brief Title: Assessment of Primary and Metastatic Brain Tumor Hypoxia With Fluoromisonidazole, FDG and Water
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI retired, study closed
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI44704
Record Dates: First submitted 2010-11-01; First posted 2010-11-23 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Brain Cancer
Keywords: brain, cancer,glioblastoma multiforme, meningioma, glioma
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Glioblastoma; Meningioma; Glioma | interventions — Fluorodeoxyglucose F18; fluoromisonidazole; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All enrolled participants will complete three imaging sessions on separate days, beginning with a research MRI, then a PET scan with FDG and [15O]water, and a PET scan with FMISO. The two PET scans will be in any order on different days within one week of each other, and preferably on consecutive days. The research MRI will be within 14 days of the first PET scan.
  Interventions: Drug: [18F]fluoro-2-deoxy-D-glucose (FDG); Drug: 1H-1-(3-[18F]-fluoro-2-hydroxy-propyl)-2-nitro-imidazole [18F]-fluoromisonidazole; Drug: [15O]water; Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: [18F]fluoro-2-deoxy-D-glucose (FDG) — Brain scan with imaging tracer used for measuring glucose metabolism in the assessment, diagnosis, and staging of patients with cancer
  Other Names: FDG; [18F]FDG; FDG-PET/CT
Drug: 1H-1-(3-[18F]-fluoro-2-hydroxy-propyl)-2-nitro-imidazole [18F]-fluoromisonidazole — Brain scan with radiopharmaceutical imaging tracer that directly assesses tumor hypoxia
  Other Names: [18F]FMISO; FMISO; FMISO-PET/CT
Drug: [15O]water — Brain scan with imaging tracer used for measuring tumor blood flow/perfusion
  Other Names: H2[15O]; H2[15O]-PET-CT
Diagnostic Test: Magnetic Resonance Imaging — Brain scan to assess tumor size and tumor blood flow/perfusion
  Other Names: MRI

SUMMARY:
Purpose of Study This exploratory clinical study will investigate FMISO (fluoromisonidazole) in patients with (1) newly diagnosed primary malignant brain tumors (WHO [World Health Organization] Grade III or IV glial-based tumors) who have not had a complete surgical resection and by contrast MRI (Magnetic resonance imaging) have residual tumor > 1.0 cm in diameter and will be receiving radiotherapy or (2) newly diagnosed brain metastasis (> 1.0 cm in diameter who will be receiving radiotherapy. The ability to accurately assess tumor hypoxia and accurately determine the amount/degree of tumor hypoxia could potentially change patient management once validated as tumor hypoxia is known to be associated with a poor prognosis [Eyler 2008].

DETAILED DESCRIPTION:
Malignant Brain Tumors (Primary and Metastatic) Despite significant advances in the understanding of brain tumor biology and genetics as well as improvements in surgical techniques, radiotherapy administration, and chemotherapy methods, many brain tumors remain incurable. Many brain tumors are highly infiltrative neoplasms, and are therefore unlikely to be cured by local treatments such as surgery, focal radiotherapy, radiosurgery or brachytherapy.

Rationale and Goals of Study The preliminary efficacy of the radiopharmaceutical, 1H-1-(3-[18F]-fluoro-2-hydroxy-propyl)-2-nitro-imidazole [18F]-fluoromisonidazole, [18F]FMISO, FMISO (fluoromisonidazole), a radiopharmaceutical that directly assess tumor hypoxia using Positron Emission Tomography(PET) will be assessed.

This preliminary/exploratory clinical study will investigate [F-18]FMISO in 30 evaluable patients with newly diagnosed primary brain tumor or brain metastasis. We expect that up to 35 -40 total patients may be enrolled in this study. This will assure that 30 evaluable patients (patients who have complete imaging results and blood metabolism data available for data analysis). In certain patients the blood metabolism data is not acceptable for final analysis typically due to difficulty in drawing it rapidly enough due to the vein collapsing during the rapid sampling required.

When possible we will also correlate FMISO uptake with the typical in-vitro test used to assess proliferation, Ki-67 (protein) and other experimental assessments of hypoxia. This correlation will be made whenever possible in those patients where tumor tissue is obtained as part of standard care.

OBJECTIVES:

Primary Objective of Study - Synopsis The primary objective of this study is to determine the association of FMISO PET (positron emission tomography) uptake (hypoxic volume (HV)), highest tumor:blood ratio [T/Bmax]), FDG ([18F]-2 fluoro-2-deoxy-d-glucose) uptake, and tumor blood flow/perfusion determined with water (H2O) and MRI and correlate these variables with overall survival (OS) and time to progression (TTP) in participants with newly diagnosed primary brain tumors or brain metastases.

The Hypotheses to be Tested

Three exploratory hypotheses will be studied. These include:

1. The first hypothesis to be tested is that increased FMISO PET uptake (hypoxic volume [HV], highest tumor:blood ratio [T/Bmax]) is correlated with a shorter overall survival and a shorter time to progression. An exploratory evaluation assessing combinations of PET imaging variables such as hypoxic volume [HV], highest tumor:blood ratio [T/Bmax], FDG-standardized uptake value (SUV), FDG quantitative parameters and blood flow as well as magnetic resonance (MR) perfusion and blood volume will be assessed to see if they correlate with survival and time to progression.
2. A second hypothesis to be tested is that FMISO is safe and non toxic in the dose administered in this study in patients with primary and metastatic brain tumors. This will be assessed in the first 10 patients enrolled in the study. Even though there have been numerous published studies using FMISO in humans in several different tumor types little human safety data has been published. Laboratory tests (except urinalysis) will be repeated at approximately 24 hours in the first 10 and compared to the screening values.
3. A third exploratory hypothesis to be tested is that FMISO uptake (hypoxic volume [HV], highest tumor:blood ratio [T/Bmax]) will correlate with increased FDG uptake and possibly with reduced blood flow/perfusion as determined with H215O PET imaging and MRI

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients. The patient must have a newly diagnosed primary malignant brain tumors (WHO Grade III or IV glial-based tumors) and not have had a complete surgical resection and by contrast MRI (obtained within 14 days prior to the FMISO study)
2. Patients must be 18 years or older for inclusion in this research study.
3. Patients must document their willingness to be followed until death or time of progression.
4. All patients must sign a written informed consent and HIPAA authorization in accordance with institutional guidelines.
5. Female patients who are not postmenopausal or surgically sterile will undergo a serum pregnancy test prior to the research PET scans.
6. Pre-treatment laboratory tests for patients receiving [18F]FMISO must be performed within 21 days prior to study entry.

Exclusion Criteria:

1. Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals.
2. Patients who are pregnant or lactating or who suspect they might be pregnant.
3. Adult patients who require monitored anesthesia for PET scanning.
4. Patients who are too claustrophobic to undergo MRI or PET imaging
5. Patients who cannot undergo MRI imaging due to MRI exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2014-05-03 (Actual); Study Completion 2014-05-03 (Actual)

PRIMARY OUTCOMES:
Determination of multi-tracer update times as related to overall survival and time to progression | estimated 2 years
  determine the association of FMISO PET uptake (hypoxic volume [HV]), highest tumor:blood ratio [T/Bmax]), FDG uptake, and tumor blood flow/perfusion determined with H215O and MRI and correlate these variables with overall survival (OS) and time to progression (TTP) in participants with newly diagnosed primary brain tumors or brain metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yap, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States